CLINICAL TRIAL: NCT02720523
Title: A Phase 2b/3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) to Placebo in Japanese Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Are on a Stable Dose of Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) and Have an Inadequate Response to csDMARDs
Brief Title: A Study to Compare Upadacitinib (ABT-494) to Placebo in Adults With Rheumatoid Arthritis (RA) Who Are on a Stable Dose of Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) and Have an Inadequate Response to csDMARDs
Acronym: SELECTSUNRISE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-663
Record Dates: First submitted 2016-03-22; First posted 2016-03-28 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; ABT-494; Japanese; Antirheumatic agents
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo / Upadacitinib 7.5 mg (Experimental): Period 1: Participants will receive placebo once daily for 12 weeks.
  Period 2: Participants will receive Upadacitinib 7.5 mg once daily for 248 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Placebo / Upadacitinib 15 mg (Experimental): Period 1: Participants will receive placebo once daily for 12 weeks.
  Period 2: Participants will receive upadacitinib 15 mg once daily for 248 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Placebo / Upadacitinib 30 mg (Experimental): Period 1: Participants will receive placebo once daily for 12 weeks.
  Period 2: Participants will receive upadacitinib 30 mg once daily until regulatory approval of RA indication in Japan at which point they will switch to receive upadacitinib 15 mg once daily. Participants will receive upadacitinib for 248 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Upadacitinib 7.5 mg / Upadacitinib 7.5 mg (Experimental): Period 1: Participants will receive upadacitinib 7.5 mg once daily for 12 weeks.
  Period 2: Participants will receive upadacitinib 7.5 mg once daily for 248 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 15 mg / Upadacitinib 15 mg (Experimental): Period 1: Participants will receive upadacitinib 15 mg once daily for 12 weeks.
  Period 2: Participants will receive upadacitinib 15 mg once daily for 248 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 30 mg / Upadacitinib 30 mg (Experimental): Period 1: Participants will receive upadacitinib 30 mg once daily for 12 weeks.
  Period 2: Participants will receive upadacitinib 30 mg once daily until regulatory approval of RA indication in Japan at which point they will switch to receive upadacitinib 15 mg once daily. Participants will receive upadacitinib for 248 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablet; Oral
  Arms: Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg; Placebo / Upadacitinib 7.5 mg
Drug: Upadacitinib — Tablet; Oral
  Other Names: ABT-494; RINVOQ™

SUMMARY:
This is a randomized, double-blind study comparing ABT-494 to placebo in Japanese participants with moderately to severely active rheumatoid arthritis who are on a stable dose of conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) and have an inadequate response.

Following marketing approval of upadacitinib for rheumatoid arthritis in Japan, this study will become a post-marketing clinical study and include a long-term extension period.

DETAILED DESCRIPTION:
This study consisted of a 35-day screening period; a 12-week randomized, double-blind, parallel-group, placebo-controlled treatment period (Period 1); a 248-week blinded long-term extension period (Period 2); and a 30-day follow-up period (call or visit).

Participants who met eligibility criteria were randomized in a 3:3:3:1:1:1 ratio to one of six treatment groups:

* Group 1: Upadacitinib 7.5 mg QD (Period 1) → upadacitinib 7.5 mg QD (Period 2)
* Group 2: Upadacitinib 15 mg QD (Period 1) → upadacitinib 15 mg QD (Period 2)
* Group 3: Upadacitinib 30 mg QD (Period 1) → upadacitinib 30 mg QD (Period 2)
* Group 4: Placebo (Period 1) → upadacitinib 7.5 mg QD (Period 2)
* Group 5: Placebo (Period 1) → upadacitinib 15 mg QD (Period 2)
* Group 6: Placebo (Period 1) → upadacitinib 30 mg QD (Period 2)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) for >= 3 months who also fulfill the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA.
* Subjects have been receiving conventional synthetic disease-modifying anti-rheumatic drug (csDMARD) therapy >= 3 months and on a stable dose for >= 4 weeks prior to the first dose of study drug.
* Subject has >= 6 swollen joints (based on 66 joint counts) and >= 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
* Subjects with prior exposure to at most one biological disease-modifying anti-rheumatic drug (bDMARD) may be enrolled (up to 20% of total number of subjects) after the required washout period. Specifically, prior to enrollment:

  1. Subjects with limited exposure to bDMARD (< 3 months) OR
  2. Subjects who are responding to bDMARD therapy but had to discontinue due to intolerability (regardless of treatment duration).

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor
* Subjects who are considered inadequate responders (lack of efficacy) to bDMARD therapy, after minimum 3 months treatment, as determined by the Investigator.
* History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis [SpA] including ankylosing spondylitis and non-radiographic axial SpA, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [currently with active symptoms]). Current diagnosis of secondary Sjogren's Syndrome is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (50):
- Japan (50):
  - Nagoya University Hospital /ID# 148005, Nagoya, Aichi-ken
  - Hamanomachi Hospital /ID# 147991, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 148008, Fukuoka, Fukuoka
  - Inoue Hospital /ID# 147966, Takasaki, Gunma
  - National Hospital Organization Asahikawa Medical Center /ID# 147994, Asahikawa, Hokkaido
  - Katayama Orthopedic Rheumatology Clinic /ID# 147976, Asahikawa, Hokkaido
  - The Hospital of Hyogo College of Medicine /ID# 147978, Nishinomiya-shi, Hyōgo
  - National Hospital Organization Sagamihara National Hospital /ID# 148221, Sagamihara-shi, Kanagawa
  - NHO Osaka Minami Med Ctr /ID# 147986, Osaka, Kawachinagano-shi
  - Kumamoto Orthopaedic Hospital /ID# 147972, Kumamoto, Kumamoto
  - Tohoku University Hospital /ID# 148435, Sendai, Miyagi
  - Medical Corporation Keiai Kai Clinic /ID# 147975, Miyazaki, Miyazaki
  - Nagaoka Red Cross Hospital /ID# 147974, Nagaoka-shi, Niigata
  - Niigata Rheumatic Center /ID# 148002, Shibata-shi, Niigata
  - Saitama Medical Center, Saitama Medical University /ID# 147965, Kawagoe-shi, Saitama
  - Jichi Medical University Hospital /ID# 148220, Shimotsuke-shi, Tochigi
  - St.Luke's International Hospital /ID# 147969, Chuo-ku, Tokyo
  - Ichinomiya Municipal Hospital /ID# 147992, Ichinomiya-shi, Tokyo
  - Toho University Ohashi Medical Center /ID# 148003, Meguro-ku, Tokyo
  - Setagaya Rheumatic Clinic /ID# 148009, Setagaya-ku, Tokyo
  - Keio University Hospital /ID# 147982, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 148007, Shinjuku-ku, Tokyo
  - Medical Corporation Uchida Clinic /ID# 148219, Sumida-ku, Tokyo
  - Tokito Clinic Rheumatology and Orthopaedics Surgery /ID# 147980, Shimonoseki-shi, Yamaguchi
  - NHO Chiba-East-Hospital /ID# 147996, Chiba
  - Sugimoto Rheumatology and Internal Medicine Clinic /ID# 147989, Fukui
  - Hopsital of the University of Occupational and Enviromental Health /ID# 147970, Fukuoka
  - Shono Rheumatism Clinic /ID# 147971, Fukuoka
  - Hiroshima Rheumatology Clinic /ID# 147981, Hiroshima
  - Matsubara Mayflower Hospital /ID# 147967, Katō
  - Kumamoto Rheumatology Clinic /ID# 147988, Kumamoto
  - St. Mary's Hospital /ID# 147979, Kurume
  - Kagawa University Hospital /ID# 148001, Kyoto
  - Marunouchi Hospital /ID# 147973, Matsumoto
  - Yu Family Clinic /ID# 147990, Miyagi
  - JP Red Cross Nagoya Daiichi /ID# 147995, Nagoya
  - Kondo Clinic for Ortho & Rheum /ID# 147984, Nagoya
  - Okayama City Gen Med Ctr /ID# 148000, Okayama
  - Oribe Clinic of Rheumatology and Internal Medicine /ID# 149308, Ōita
  - Miyashita Rheumatology Clinic /ID# 147997, Ōmura
  - Sagawa Akira Rheumatology Clin /ID# 147987, Sapporo
  - Sapporo City General Hospital /ID# 147968, Sapporo
  - Hikarigaoka Spellman Hospital /ID# 147993, Sendai
  - Honjo Rheumatism Clinic /ID# 147983, Takaoka
  - Takikawa Municipal Hospital /ID# 149309, Takikawa
  - Juntendo University Hospital /ID# 147999, Tokyo
  - National Hospital Organization Tokyo Medical Center /ID# 147998, Tokyo
  - Nihon University Itabashi Hosp /ID# 147977, Tokyo
  - Oki Medical Clinic /ID# 147985, Tomakomai
  - Toneyama National Hospital /ID# 148006, Toyonaka

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Kameda H, Takeuchi T, Yamaoka K, Oribe M, Kawano M, Zhou Y, Othman AA, Pangan AL, Kitamura S, Meerwein S, Tanaka Y. Efficacy and safety of upadacitinib in Japanese patients with rheumatoid arthritis (SELECT-SUNRISE): a placebo-controlled phase IIb/III study. Rheumatology (Oxford). 2020 Nov 1;59(11):3303-3313. doi: 10.1093/rheumatology/keaa084. PMID 32277824
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Kameda H, Takeuchi T, Yamaoka K, Oribe M, Kawano M, Yokoyama M, Pangan AL, Konishi Y, Meerwein S, Tanaka Y. Efficacy and safety of upadacitinib over 84 weeks in Japanese patients with rheumatoid arthritis (SELECT-SUNRISE). Arthritis Res Ther. 2021 Jan 6;23(1):9. doi: 10.1186/s13075-020-02387-6. PMID 33407801
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M14-663#additional-resources-section

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with active rheumatoid arthritis (RA) and an inadequate response to conventional synthetic disease-modifying anti-rheumatic drug (csDMARDs) were enrolled at 49 sites in Japan.
  The study is currently ongoing, results are reported up to Week 60, as of the data cutoff date of 12 July 2018.
Pre-assignment Details: Participants were randomized to 1 of 3 doses of upadacitinib or placebo in Period 1. Participants who completed week 12 could continue in the study; participants in the upadacitinib groups continued on the same dose of upadacitinib, participants in the placebo group switched to upadacitinib 7.5, 15, or 30 mg per the pre-specified randomization.
Groups:
- Period 1: Placebo: Participants randomized to receive placebo once daily (QD) for 12 weeks in Period 1.
- Period 1: Upadacitinib 7.5 mg: Participants randomized to receive upadacitinib 7.5 mg once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily for 12 weeks in Period 1.
- Period 2: Upadacitinib 7.5 mg: Participants received upadacitinib 7.5 mg QD from Week 12 to Week 260 during the long-term extension period.
- Period 2: Upadacitinib 15 mg: Participants received upadacitinib 15 mg QD from Week 12 to Week 260 during the long-term extension period.
- Period 2: Upadacitinib 30 mg: Participants received upadacitinib 30 mg QD from Week 12 to Week 260 during the long-term extension period.
Period: Period 1: Placebo-controlled Period
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 7.5 mg | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 2: Upadacitinib 7.5 mg | Period 2: Upadacitinib 15 mg | Period 2: Upadacitinib 30 mg
Started | 49 | 49 | 49 | 50 | 0 | 0 | 0
Completed | 47 | 49 | 47 | 44 | 0 | 0 | 0
Not Completed | 2 | 0 | 2 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Period 2: Long-term Extension Period
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 7.5 mg | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 2: Upadacitinib 7.5 mg | Period 2: Upadacitinib 15 mg | Period 2: Upadacitinib 30 mg
Started | 0 | 0 | 0 | 0 | 65 (Includes participants originally randomized to placebo and upadacitinib 7.5 mg) | 62 (Includes participants originally randomized to placebo and upadacitinib 15 mg) | 60 (Includes participants originally randomized to placebo and upadacitinib 30 mg)
Completed (Completed study as of the data cutoff date of 12 July 2018) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 65 | 62 | 60
Not completed — Ongoing | 0 | 0 | 0 | 0 | 57 | 54 | 45
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 7 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Participants randomized to receive placebo once daily for 12 weeks in Period 1.
- Upadacitinib 7.5 mg: Participants randomized to receive upadacitinib 7.5 mg once daily for 12 weeks in Period 1.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily for 12 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 49 | 49 | 49 | 50 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.04) | 55.8 (11.02) | 56.0 (12.50) | 54.7 (12.22) | 55.2 (12.14)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 7 | 5 | 8 | 3 | 23
  45 to < 65 years | 31 | 32 | 30 | 34 | 127
  ≥ 65 years | 11 | 12 | 11 | 13 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 36 | 43 | 155
  Male | 7 | 15 | 13 | 7 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 49 | 49 | 49 | 50 | 197
Duration of RA Diagnosis [Mean (Standard Deviation); unit: years] | 4.8 (4.86) | 6.7 (7.15) | 5.9 (7.20) | 4.5 (4.30) | 5.5 (6.03)
Prior Biological Disease-modifying Anti-rheumatic Drug (bDMARD) Use [Count of Participants; unit: Participants]
  Yes | 3 | 5 | 6 | 3 | 17
  No | 46 | 44 | 43 | 47 | 180
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  joints | 16.8 (11.42) | 16.3 (8.89) | 17.8 (12.58) | 16.3 (10.79) | 16.8 (10.93)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  joints | 10.9 (4.65) | 11.7 (4.89) | 14.0 (7.82) | 11.7 (5.32) | 12.1 (5.88)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain."
  mm | 56.1 (20.83) | 57.8 (22.62) | 50.5 (25.41) | 45.5 (21.85) | 52.4 (23.09)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity.
  mm | 53.8 (21.72) | 59.0 (22.51) | 49.3 (24.89) | 47.8 (22.79) | 52.4 (23.25)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 49 | 49 | 48 | 50 | 196
    (all) | 57.4 (18.62) | 55.6 (16.65) | 58.8 (20.21) | 57.6 (21.38) | 57.4 (19.19)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  units on a scale | 1.0 (0.67) | 0.9 (0.67) | 1.0 (0.67) | 0.9 (0.60) | 0.9 (0.65)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 17.9 (20.53) | 13.3 (12.80) | 15.8 (18.23) | 12.4 (13.67) | 14.8 (16.62)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 42.9 [29.0 to 56.7] | 75.5 [63.5 to 87.6] | 83.7 [73.3 to 94.0] | 80.0 [68.9 to 91.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 32.7, 95% CI 2-sided [14.3 to 51.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 40.8, 95% CI 2-sided [23.5 to 58.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 37.1, 95% CI 2-sided [19.4 to 54.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 4: Comparison: Upadacitinib 7.5 mg vs Upadacitinib 15 mg vs Upadacitinib 30 mg; Test type: Other — Cochran-Armitage test was conducted for demonstrating a dose response relationship; p < 0.001, Cochran-Armitage test

2. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28) (CRP) at Week 12
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Baseline and Week 12
Population: Full analysis set; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
scores on a scale | -0.79 [-1.158 to -0.426] | -2.08 [-2.430 to -1.727] | -2.39 [-2.735 to -2.043] | -2.41 [-2.776 to -2.050]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model including treatment as the fixed factor, and baseline value and the stratification factor prior bDMARD use as covariates; Least Squares (LS) Mean Difference = -1.29, 95% CI 2-sided [-1.693 to -0.880] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.60, 95% CI 2-sided [-2.005 to -1.190] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 2, analysis 1]; LS Mean Difference = -1.62, 95% CI 2-sided [-2.027 to -1.216] — Difference = Upadacitinib - Placebo

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
scores on a scale | -0.10 [-0.245 to 0.043] | -0.41 [-0.545 to -0.267] | -0.45 [-0.583 to -0.309] | -0.49 [-0.636 to -0.347]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA model includes treatment as the fixed factor, and the baseline value and stratification factor prior bDMARD use as the covariates; LS Mean Difference = -0.30, 95% CI 2-sided [-0.465 to -0.144] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -0.34, 95% CI 2-sided [-0.505 to -0.184] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -0.39, 95% CI 2-sided [-0.550 to -0.229] — Difference = Upadacitinib - Placebo

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 16.3 [6.0 to 26.7] | 40.8 [27.1 to 54.6] | 65.3 [52.0 to 78.6] | 58.0 [44.3 to 71.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 24.5, 95% CI 2-sided [7.3 to 41.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 49.0, 95% CI 2-sided [32.1 to 65.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 41.7, 95% CI 2-sided [24.5 to 58.8] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 2.0 [0.0 to 6.0] | 20.4 [9.1 to 31.7] | 34.7 [21.4 to 48.0] | 28.0 [15.6 to 40.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 18.4, 95% CI 2-sided [6.4 to 30.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 32.7, 95% CI 2-sided [18.7 to 46.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 26.0, 95% CI 2-sided [12.9 to 39.0] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 47 | 49 | 48 | 44
scores on a scale | 2.88 [1.03 to 4.72] | 7.21 [5.43 to 8.99] | 6.38 [4.60 to 8.15] | 8.81 [6.93 to 10.68]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; MMRM model with fixed effects of treatment, visit and treatment-by-visit interaction, prior bDMARD use, and baseline value as covariate; LS Mean Difference = 4.33, 95% CI 2-sided [2.10 to 6.57] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p = 0.002, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 3.50, 95% CI 2-sided [1.25 to 5.75] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 5.93, 95% CI 2-sided [3.64 to 8.22] — Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12
Description: Low disease activity. was defined as a DAS28 score less than or equal to 3.2. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 18.4 [7.5 to 29.2] | 53.1 [39.1 to 67.0] | 69.4 [56.5 to 82.3] | 72.0 [59.6 to 84.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 34.7, 95% CI 2-sided [17.0 to 52.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 51.0, 95% CI 2-sided [34.2 to 67.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 53.6, 95% CI 2-sided [37.1 to 70.1] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 12
Description: Clinical remission was defined as a DAS28 (CRP) score less than 2.6. The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 6.1 [0.0 to 12.8] | 36.7 [23.2 to 50.2] | 57.1 [43.3 to 71.0] | 50.0 [36.1 to 63.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 30.6, 95% CI 2-sided [15.5 to 45.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 51.0, 95% CI 2-sided [35.6 to 66.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 43.9, 95% CI 2-sided [28.5 to 59.3] — Response Rate Difference = Upadacitinib - Placebo

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 1
Description: as for outcome 1
Time Frame: Baseline and Week 1
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 1 or for whom ACR data were missing at Week 1 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 49 | 49 | 49 | 50
percentage of participants | 8.2 [0.5 to 15.8] | 30.6 [17.7 to 43.5] | 24.5 [12.4 to 36.5] | 34.0 [20.9 to 47.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 22.4, 95% CI 2-sided [7.4 to 37.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p = 0.026, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 16.3, 95% CI 2-sided [2.1 to 30.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factor prior bDMARD use; Response Rate Difference = 25.8, 95% CI 2-sided [10.6 to 41.0] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Change From Baseline in in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) at Week 12
Description: The FACIT Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a four point Likert scale. The FACIT Fatigue Scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 47 | 49 | 48 | 44
scores on a scale | 1.81 [-0.35 to 3.97] | 4.47 [2.38 to 6.55] | 3.60 [1.53 to 5.68] | 2.66 [0.48 to 4.85]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.040, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 2.66, 95% CI 2-sided [0.12 to 5.20] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p = 0.169, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 1.79, 95% CI 2-sided [-0.77 to 4.35] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p = 0.516, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = 0.85, 95% CI 2-sided [-1.73 to 3.43] — Difference = Upadacitinib - Placebo

11. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Work Instability Scale (RA-WIS) at Week 12
Description: RA-WIS is a simple validated tool to evaluate work instability (the consequence of a mismatch between an individual's functional ability and their work tasks). RA-WIS consists of 23 questions relating to the participant's functioning in their work environment, each answered as Yes or No. The total score is the number of questions answered Yes, and ranges from 0 to 23.
  A score < 10 means low risk and no action is needed, scores between 10 and 17 indicate medium risk and appropriate advice and information should be given. If the score is > 17, it means high risk and it could warrant referral.
  A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants who were working and with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 34 | 31 | 24 | 18
scores on a scale | -0.69 [-2.58 to 1.21] | -3.22 [-5.09 to -1.36] | -2.74 [-4.75 to -0.74] | -2.24 [-4.40 to -0.09]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.021, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -2.54, 95% CI 2-sided [-4.68 to -0.39] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p = 0.080, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -2.06, 95% CI 2-sided [-4.36 to 0.25] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p = 0.220, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.56, 95% CI 2-sided [-4.06 to 0.94] — Difference = Upadacitinib - Placebo

12. Secondary Outcome: Change From Baseline in the Severity of Morning Stiffness at Week 12
Description: Morning stiffness severity was determined by the Patient's Assessment of Severity and Duration of Morning Stiffness questionnaire. Participants rated the severity of morning stiffness on awakening over the past 7 days on a scale from 0 (No morning stiffness) to 10 (Worst possible morning stiffness).
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 47 | 49 | 48 | 44
scores on a scale | -1.02 [-1.65 to -0.39] | -2.83 [-3.44 to -2.22] | -2.84 [-3.45 to -2.23] | -2.98 [-3.62 to -2.34]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.81, 95% CI 2-sided [-2.57 to -1.04] — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.82, 95% CI 2-sided [-2.59 to -1.05] — Difference = Upadacitinib - Placebo
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.96, 95% CI 2-sided [-2.73 to -1.18] — Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: Period 1: Weeks 1 to 12; Period 2: Weeks 12 to 60
Groups:
- Period 1: Placebo: Participants received placebo once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 7.5 mg: Participants received upadacitinib 7.5 mg once daily for 12 weeks in Period 1
- Period 1: Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 12 weeks in Period 1
- Period 1: Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 12 weeks in Period 1.
- Period 1+2: Upadacitinib 7.5 mg: Participants originally randomized to upadacitinib 7.5 mg received upadacitinib 7.5 mg once daily for 12 weeks in Period 1 and up to Week 60 in Period 2. Participants originally randomized to placebo received upadacitinib 7.5 mg from Week 12 to Week 60.
- Period 1+2: Upadacitinib 15 mg: Participants originally randomized to upadacitinib 15 mg received upadacitinib 15 mg once daily for 12 weeks in Period 1 and up to Week 60 in Period 2. Participants originally randomized to placebo received upadacitinib 15 mg from Week 12 to Week 60.
- Period 1+2: Upadacitinib 30 mg: Participants originally randomized to upadacitinib 30 mg received upadacitinib 30 mg once daily for 12 weeks in Period 1 and up to Week 60 in Period 2. Participants originally randomized to placebo received upadacitinib 30 mg from Week 12 to Week 60.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 7.5 mg | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 1+2: Upadacitinib 7.5 mg | Period 1+2: Upadacitinib 15 mg | Period 1+2: Upadacitinib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/50 | 0/65 | 0/64 | 2/66
Serious Adverse Events (participants affected / at risk) | 0/49 | 1/49 | 1/49 | 5/50 | 9/65 | 14/64 | 18/66
Other Adverse Events (participants affected / at risk) | 11/49 | 20/49 | 15/49 | 27/50 | 55/65 | 55/64 | 60/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=49) | Period 1: Upadacitinib 7.5 mg (N=49) | Period 1: Upadacitinib 15 mg (N=49) | Period 1: Upadacitinib 30 mg (N=50) | Period 1+2: Upadacitinib 7.5 mg (N=65) | Period 1+2: Upadacitinib 15 mg (N=64) | Period 1+2: Upadacitinib 30 mg (N=66)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Philadelphia chromosome positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=49) | Period 1: Upadacitinib 7.5 mg (N=49) | Period 1: Upadacitinib 15 mg (N=49) | Period 1: Upadacitinib 30 mg (N=50) | Period 1+2: Upadacitinib 7.5 mg (N=65) | Period 1+2: Upadacitinib 15 mg (N=64) | Period 1+2: Upadacitinib 30 mg (N=66)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (8)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 10 (10)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 8 (8) | 2 (2) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 13 (17) | 6 (8) | 5 (5)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 5 (7)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (7) | 4 (5) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 4 (8)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 4 (5) | 5 (5)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 9 (9) | 10 (10)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 9 (10) | 6 (6)
Nasopharyngitis (Infections and infestations) | 5 (8) | 5 (6) | 6 (6) | 9 (11) | 35 (71) | 35 (59) | 29 (64)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 5 (6) | 5 (5)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (2) | 4 (5)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 7 (8) | 8 (11)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 6 (8) | 4 (4)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 6 (8)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 4 (6)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 5 (6) | 7 (10)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 7 (7)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 8 (8) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02720523/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT02720523/SAP_001.pdf